CLINICAL TRIAL: NCT07181642
Title: Efficacy of a Diaphragmatic Breathing Program in Adults With Sleep Bruxism: A Randomized Controlled Trial
Brief Title: Diaphragmatic Breathing for Sleep Bruxism in Adults: A Randomized Controlled Trial
Acronym: DB4SB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Chtioui Hajer, Assistant, Removable Partial Dentures, University of Monastir
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DB-SB-RCT-2025
Record Dates: First submitted 2025-09-11; First posted 2025-09-18 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Bruxism; Bruxism, Sleep-Related
MeSH Terms: conditions — Bruxism; Sleep Bruxism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group - Diaphragmatic Breathing (Experimental): Participants will learn and practice diaphragmatic breathing exercises daily for 4 weeks.
  Interventions: Behavioral: Diaphragmatic Breathing Program
- Placebo Group (Placebo Comparator): Participants will listen to neutral music of the same duration before sleep. This activity does not include any therapeutic breathing exercises and is intended as a control.
  Interventions: Behavioral: Neutral Music Listening

INTERVENTIONS:
Behavioral: Diaphragmatic Breathing Program — Participants will learn diaphragmatic breathing exercises and practice them daily for 4 weeks before bedtime.
  Other Names: Deep Breathing Exercises
  Arms: Experimental Group - Diaphragmatic Breathing
Behavioral: Neutral Music Listening — Participants will listen to neutral music of the same duration before sleep. This activity does not include any therapeutic breathing exercises and is intended as a control
  Other Names: placebo
  Arms: Placebo Group

SUMMARY:
The goal of this clinical trial is to learn if a diaphragmatic breathing program can reduce sleep bruxism in adults. The main questions it aims to answer are:

Can diaphragmatic breathing lower the frequency of teeth grinding during sleep?

Can it reduce jaw discomfort and improve sleep quality?

Participants will:

Attend sessions to learn diaphragmatic breathing exercises

Practice these exercises daily at home for 4 weeks

Complete questionnaires and clinical assessments before and after the program

Participation is safe, with minimal risks, such as mild fatigue during exercises. The study will help determine if diaphragmatic breathing is an effective way to manage sleep bruxism

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed sleep bruxism
* Provision of consent

Exclusion Criteria:

* • Current use of medications affecting sleep or neuromuscular function

  * History of severe neurological or psychiatric disorders
  * Ongoing use of a dental reconditioning splint or occlusal device
  * Inability to informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2025-09-15 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-11-14 (Actual)

PRIMARY OUTCOMES:
Sleep Bruxism Frequency | 4 weeks
  The frequency of sleep bruxism episodes will be assessed using the standardized STAB questionnaire and patient self-reports. Measurements will be taken at baseline (before starting the intervention) and at the end of the 4-week program to determine any change in bruxism frequency.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Habib Bougatfa Bizerte, Bizerte, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided